CLINICAL TRIAL: NCT01060202
Title: A Prospective, Open-label, Multicenter Observational Study to Evaluate the QoL of Non-transplant Candidate Multiple Myeloma Patients Treated With Early Bortezomib
Brief Title: Quality of Life of Non-transplant Candidate Multiple Myeloma Patients Treated With Early Bortezomib
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR016750; BOR-KOR-5022 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Bortezomib; Velcade; QoL; Proteasome inhibitor; EORTC QLQ C30; EQ 5D
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bortezomib
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — This is an observational study. Patients receiving bortezomib injection intravenously (into a vein) 1.3 mg/m2 twice a week for 21 days will be observed.

SUMMARY:
This study will observe the degree of the quality of life in non-transplant candidate patients with multiple myeloma before and after bortezomib administration by using EORTC-QLQ C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core30) and EQ-5D (EuroQol-5 Dimensions). Both tools are validated research instruments used to measure the quality of life in cancer patients and consequently will provide fundamental data regarding the quality of life in patients with multiple myeloma by analyzing factors that affect the quality of life.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a plasma cell malignancy with progression marked by symptoms and signs of lowered resistance to infection, skeletal destruction, renal failure, and anemia. It is incurable and follows a relapsing course, with a median survival of approximately 4-5 years. The various therapies associated with disease control, are often associated with significant side effects, and ultimately, patients relapse. Therefore, assessment of health-related quality of life (HRQL) represents an important tool for evaluating the value of effective therapies when weighed against the potential toxic effects of treatment from the patient's perspective. Patients diagnosed with MM suffer from pain, fatigue, reduced physical and role functioning, and reduced overall HRQL compared with an age- and gender-matched population. These symptoms can improve with successful treatment with either cytotoxic therapy or supportive care. Many clinical studies for the treatment of multiple myeloma have been conducted in Korea, but none of them have evaluated the improvement in the quality of life in patients with multiple myeloma. Most study variables used to evaluate the quality of life of patients with multiple myeloma are subjective and limited. This study will observe the degree of the quality of life of patients in the early status of multiple myeloma before and after bortezomib administration by using EORTC-C30 (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core30) and EQ-5D (EuroQol-5 Dimensions), validated research instruments used to measure the quality of life in cancer patients and consequently will provide fundamental data regarding the quality of life in patients with multiple myeloma. Observational Study - No investigational drug administered.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic multiple myeloma patient
* ECOG score less than 3
* Patient is not a candidate for stem cell transplantation
* Previous treatment duration is less than 6 months
* Previous treatment response is less than partial response (PR)
* Willing and able to complete the questionnaire
* Patients (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Known hypersensitivity to bortezomib
* Acute severe infection requiring antibiotics therapy
* Pre-existing peripheral neuropathy greater than or equal to grade 2
* Uncontrolled or severe cardiovascular disease
* Pregnancy or breastfeeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-transplant candidate patients who are newly prescribed bortezomib injection as a secondary agent for the treatment of multiple myeloma, those of whom can understand and fill out questionnaire, and agree to provide information will be included.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2009-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The change in the quality of life as measured by EORTC QLQ-C30 and EQ-5D before and after the administration of bortezomib | On day 1 at the first cycle, 12 weeks, 24 weeks

SECONDARY OUTCOMES:
Relationship between the primary outcome and the complete remission (CR) rate | 12 weeks and 24 weeks
Relationship between the primary outcome and overall response | 12 weeks and 24 weeks
Relationship between the primary outcome and the time to response | 12 weeks and 24 weeks
Relationship between the primary outcome and the survival | 12 weeks and 24 weeks
Adverse events | every 3 week cycle

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea

REFERENCES:
- See also: A prospective, open-label, multicenter observational study to evaluate the QoL of nontransplant candidate multiple myeloma patients treated with the early bortezomib — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=341&filename=CR016750_CSR.pdf